CLINICAL TRIAL: NCT02040675
Title: Use of NAVA-catheter Positioning Screen to Identify Different Cardiac Arrhythmias
Status: Completed | Type: Observational
Sponsor: ProMedica Health System (Other)
Responsible Party: Principal Investigator, Howard Stein, Director Neonatology, ProMedica Health System
Other Study IDs: TCH01
Record Dates: First submitted 2014-01-13; First posted 2014-01-20 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Cardiac Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to validate a novel method of diagnosing arrhythmias using the NAVA catheter-positioning screen in patients who have a NAVA catheter in place.

DETAILED DESCRIPTION:
The population will be a convenience sample of adults with various arrhythmias who are scheduled to undergo an electrophysiology study and-or ablation (EPSA) under general anesthesia (GETA) at The Toledo Hospital.

After the patient has been successfully intubated at the beginning of the procedure, a trained nurse, using standard technique for placement of a oro/nasogastric tube, will place an appropriately sized NAVA catheter in the patient. The lumen of the NAVA tube can be used as a conventional oro/nasogastric tube and the electrodes will be connected to the Servo-I ventilator. Although the Servo-I is a ventilator, it will be used only as a monitor for this study. The position of the nasogastric tube will then be refined using the catheter positioning screen as needed.

During the course of the EPSA various arrhythmias may become evident. When these are noted, screen shots will be saved on the Servo-i monitor. Surface and electrogram recordings will be saved at the same time. The NAVA catheter will be disconnected from the Servo-I monitor during the ablation part of the procedure to prevent inadvertent damage to the monitor.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac arrhythmia

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will be a convenience sample of adults with various arrhythmias who are scheduled to undergo an electrophysiology study and-or ablation (EPSA) under general anesthesia (GETA) at The Toledo Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2014-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Types of cardiac arrhythmia | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Howard Stein, MD, Principal Investigator — Promedica Toledo CHildren's Hospital
Locations (1):
- Promedica Toledo Hospital, Toledo, Ohio, United States